CLINICAL TRIAL: NCT07346326
Title: Comparative Study of Functional Outcomes Between Peroneus Longus and Hamstring Tendon Autografts in Arthroscopic ACL Reconstruction: A Randomized Controlled Trial
Brief Title: Comparative Study of Functional Outcomes Between Peroneus Longus and Hamstring Tendon Autografts in Arthroscopic ACL Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: Khyber Medical College, Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/12
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: ACL reconstruction; Hamstring tendon autograft; Functional outcomes; Arthroscopy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two parallel groups receiving a different type of tendon autograft.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the surgical intervention, the participating surgeons and patients cannot be blinded to the group assignment. However, the independent assessor responsible for collecting the primary outcome (Lysholm Knee Score) will be blinded to which graft type the participant received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hamstring Tendon (HST) Autograft Group (Experimental): Participants will undergo arthroscopic anterior cruciate ligament (ACL) reconstruction using an autograft harvested from their own ipsilateral hamstring tendons (semitendinosus and gracilis). The tendons will be harvested, prepared as a quadrupled graft, and fixed using an Endobutton on the femoral side and an adjustable button system (ABS) on the tibial side via a standard single-bundle technique.
  Interventions: Procedure: Hamstring Tendon Autograft Harvest and ACL Reconstruction
- Peroneus Longus Tendon (PLT) Autograft Group (Active Comparator): Participants will undergo arthroscopic anterior cruciate ligament (ACL) reconstruction using an autograft harvested from their own ipsilateral peroneus longus tendon (PLT). The tendon will be harvested through a 2-3 cm incision proximal to the lateral malleolus, with a tenodesis of the peroneus brevis performed at the donor site. The graft will be prepared and fixed using an Endobutton on the femoral side and an adjustable button system (ABS) on the tibial side via a standard single-bundle technique.
  Interventions: Procedure: Peroneus Longus Tendon Autograft Harvest and ACL Reconstruction

INTERVENTIONS:
Procedure: Hamstring Tendon Autograft Harvest and ACL Reconstruction — Arthroscopic anterior cruciate ligament (ACL) reconstruction performed under spinal anesthesia, utilizing an autograft harvested from the patient's own ipsilateral semitendinosus and gracilis (hamstring) tendons. The harvested tendons are prepared as a quadrupled graft. Reconstruction follows a standard single-bundle technique with graft fixation using an Endobutton on the femoral side and an adjustable button system on the tibial side.
  Other Names: HST autograft; Quadrupled semitendinosus-gracilis autograft
  Arms: Hamstring Tendon (HST) Autograft Group
Procedure: Peroneus Longus Tendon Autograft Harvest and ACL Reconstruction — Arthroscopic anterior cruciate ligament (ACL) reconstruction performed under spinal anesthesia, utilizing an autograft harvested from the patient's own ipsilateral peroneus longus tendon (PLT). The tendon is harvested through a 2-3 cm incision proximal to the lateral malleolus, with a tenodesis of the peroneus brevis performed at the donor site. Reconstruction follows a standard single-bundle technique with graft fixation using an Endobutton on the femoral side and an adjustable button system on the tibial side.
  Arms: Peroneus Longus Tendon (PLT) Autograft Group

SUMMARY:
This is a prospective, single-blinded, randomized controlled trial. Sixty patients (≥18 years) with an isolated ACL injury will be randomly assigned to receive an ACL reconstruction using either a Peroneus Longus Tendon (PLT) autograft or a Hamstring Tendon (HST) autograft. The primary objective is to compare early functional outcomes between the two groups at 6 weeks and 3 months post-surgery, using the Lysholm Knee Score. The study aims to demonstrate the non-inferiority of the PLT graft. All surgeries will be performed arthroscopically at Khyber Teaching Hospital, Peshawar, followed by a standardized rehabilitation protocol.

DETAILED DESCRIPTION:
This study compares two autograft sources for anterior cruciate ligament (ACL) reconstruction. While the hamstring tendon (HST) is a widely used standard, it is associated with donor-site complications such as anterior knee pain and weakness. The peroneus longus tendon (PLT) has emerged as a potential alternative, offering similar biomechanical strength with the possibility of reduced donor-site morbidity. However, robust comparative data, particularly focusing on early functional recovery, remain limited, creating a need for high-quality evidence to guide surgical decision-making.

To this end, the trial is designed as a single-center, prospective, randomized controlled study. Sixty patients will be randomly assigned to receive ACL reconstruction using either a PLT or HST autograft, with functional outcomes assessed via the Lysholm Knee Score at six weeks and three months postoperatively. The methodology includes rigorous allocation concealment, blinding of the outcome assessor, and an intention-to-treat statistical analysis to robustly test the non-inferiority of the PLT graft.

The trial has received ethical approval, and all participants will provide informed consent. The findings aim to contribute meaningful evidence to clinical practice and will be disseminated through peer-reviewed publications and scientific conferences, with the goal of informing safer and more effective surgical choices for patients with ACL injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Isolated, primary Anterior Cruciate Ligament (ACL) injury confirmed by clinical assessment and Magnetic Resonance Imaging (MRI).
* Provides written informed consent for the surgical procedure and study participation, including follow-up assessments.

Exclusion Criteria:

* Multiligament knee injuries (e.g., concomitant PCL, MCL, or LCL injuries).
* Previous surgery or history of fracture in the involved lower limb.
* Radiographic evidence of osteoarthritis in the affected knee.
* Presence of any neuromuscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Knee instability | 6 weeks, 3 months after surgery
  A Lysholm Knee Score validated patient-reported outcome measure assessing knee function, symptoms, and instability. Scores range from 0 to 100, with higher scores indicating better function. Outcomes are categorized as Excellent (>90), Good (65-89), or Poor (<64).
Knee function | 6 weeks, 3 months after surgery
  A Lysholm Knee Score validated patient-reported outcome measure assessing knee function, symptoms, and instability. Scores range from 0 to 100, with higher scores indicating better function. Outcomes are categorized as Excellent (>90), Good (65-89), or Poor (<64).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Syed Dil Bagh Ali Shah, MBBS, Principal Investigator — Khyber Teaching Hospital; Dr Rao Erbaz Hassan, MBBS, Principal Investigator — Khyber Teaching Hospital; Dr Imtiaz, MBBS, Principal Investigator — Khyber Teaching Hospital
Locations (1):
- Khyber Teaching Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the primary publication will be made available to researchers upon reasonable request, following the completion of the trial and primary analysis. This includes demographic data, baseline clinical characteristics, surgical details, and outcome measures (Lysholm Knee Scores at all time points).
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Data will become available beginning 6 months after the publication of the primary results manuscript. Data will be available for a minimum of 5 years.
Access Criteria: Data access requests will be reviewed by the trial's principal investigator and steering committee. Requestors will be required to submit a methodologically sound research proposal. Access will be granted following the execution of a data use/sharing agreement that commits the requestor to: 1) using the data only for the approved research, 2) securing the data appropriately, 3) destroying the data after analyses are complete, 4) not attempting to re-identify participants, and 5) acknowledging the data source in any publications. Proposals must also obtain approval from an authorized Institutional Review Board (IRB) or Ethics Committee.

REFERENCES:
- [Background] Corry IS, Webb JM, Clingeleffer AJ, Pinczewski LA. Arthroscopic reconstruction of the anterior cruciate ligament. A comparison of patellar tendon autograft and four-strand hamstring tendon autograft. Am J Sports Med. 1999 Jul-Aug;27(4):444-54. doi: 10.1177/03635465990270040701. PMID 10424213
- [Background] Adachi N, Ochi M, Uchio Y, Sakai Y, Kuriwaka M, Fujihara A. Harvesting hamstring tendons for ACL reconstruction influences postoperative hamstring muscle performance. Arch Orthop Trauma Surg. 2003 Nov;123(9):460-5. doi: 10.1007/s00402-003-0572-2. Epub 2003 Aug 14. PMID 12920536
- [Background] Rhatomy S, Asikin AIZ, Wardani AE, Rukmoyo T, Lumban-Gaol I, Budhiparama NC. Peroneus longus autograft can be recommended as a superior graft to hamstring tendon in single-bundle ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2019 Nov;27(11):3552-3559. doi: 10.1007/s00167-019-05455-w. Epub 2019 Mar 15. PMID 30877316
- [Background] He J, Tang Q, Ernst S, Linde MA, Smolinski P, Wu S, Fu F. Peroneus longus tendon autograft has functional outcomes comparable to hamstring tendon autograft for anterior cruciate ligament reconstruction: a systematic review and meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2021 Sep;29(9):2869-2879. doi: 10.1007/s00167-020-06279-9. Epub 2020 Sep 27. PMID 32984919
- [Background] Asif N, Khan MJ, Singhal U, Anwer A, Firoz MA, Rashid M. Randomized Controlled Study Comparing Hamstring Graft and Peroneus Longus Tendon Graft in Arthroscopic ACL Reconstruction. J Orthop Case Rep. 2024 Nov;14(11):240-245. doi: 10.13107/jocr.2024.v14.i11.4980. PMID 39524299